CLINICAL TRIAL: NCT06236412
Title: Effects of Breastfeeding Education Interventions During Pregnancy on Breastfeeding Practices in Rural South Ethiopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wachemo University (Other)
Collaborators: Nestlé Foundation (Other)
Responsible Party: Principal Investigator, Belayneh Hamdela Jena, Assistant Professor of Epidemiology, Wachemo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WachemoU
Record Dates: First submitted 2024-01-11; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Pre-lacteal Feeding; Colostrum Feeding; Early Initiation of Breastfeeding; Exclusive Breastfeeding
Keywords: Breastfeeding practice; Health education; Pregnancy; Rural
MeSH Terms: conditions — Breast Feeding; Health Education

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial using a three-arm parallel group design will be implemented. A post-test only trial design. The three arms are: pregnant woman alone, pregnant woman with mother-in-law, and pregnant woman in routine care (control).
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are data collectors who will be trained for only outcome data collection. They will not be involved in any manipulations other than outcome data collection. They will not be involved in baseline data collection as well. They will not have information about which group receive the intervention and which group not. Their only purpose is to interview participants about the outcome status, which will be prepared by the investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention arm 1: pregnant woman alone (Experimental): Breastfeeding education:
  Breast milk features, contents, advantages, how to improve its quality, and quantity.
  Pre-lacteal feeding: meaning, addressing misconceptions, to avoid any foods/fluids up to 6 months and its harmful effects Colostrum feeding: meaning, its contents, advantages and addressing related misconceptions Early initiation of breastfeeding: proper time to initiation of breastfeeding & advantages for mother & child Exclusive breastfeeding: meaning, advantages, how long to exclusively breastfed.
  They will also receive iron suphate/folic acid supplementation as recommended practice, at least for 90 days (90+ days)
  Interventions: Behavioral: Health education
- Intervention arm 2: Pregnant woman with mother-in-law (Experimental): Breastfeeding education:
  Breast milk features, contents, advantages, how to improve its quality, and quantity.
  Pre-lacteal feeding: meaning, addressing misconceptions, to avoid any foods/fluids up to 6 months and its harmful effects Colostrum feeding: meaning, its contents, advantages and addressing related misconceptions Early initiation of breastfeeding: proper time to initiation of breastfeeding & advantages for mother & child Exclusive breastfeeding: meaning, advantages, how long to exclusively breastfed.
  They will also receive iron suphate/folic acid supplementation as recommended practice, at least for 90 days (90+ days)
  Interventions: Behavioral: Health education
- Control arm: 'Pregnant woman in routine care'. (Active Comparator): Pregnant women in this arm receive routine care, which includes existing community and health facility-based health care. The routine (standard) care at the community level includes those services given by the health extension workers such as hygiene (personal, food and environmental hygiene), and family health services such as antenatal care, postnatal care, immunization, breastfeeding, nutrition. In this trial, the control arm will receive counseling about antenatal care, health facility delivery, postnatal care, dietary intake (additional meal during pregnancy and after delivery), hygiene, and less deep information about breastfeeding practices such as on demand feeding day and night, exclusive breastfeeding, continuing breastfeeding for at least 24 months, to balance and make the frequency and duration with that of the intervention arm. They will also receive iron suphate/folic acid supplementation as recommended practice, at least for 90 days (90+ days)
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Health education — Health education about the contents listed under each arm will be provided for the participants.

SUMMARY:
Background: Breast milk is primary source of nutrition for newborns, containing both macro and micro nutrients. However, breastfeeding practices vary from setting-to-setting, and affect newborn's growth and development. In Ethiopia, sizable proportion of newborns (19%) do not feed colostrum; instead, pre-lacteal foods are given until colostrum is partly or fully removed. This obviously delays timely initiation, and affects exclusive breastfeeding. Furthermore, avoiding colostrum and giving pre-lacteal foods make newborns more susceptible for infections and/or diarrheal diseases that lead to death. Additionally, 26% of newborns exposed for pre-lacteal feeding, 27% initiate breastfeeding lately and 41% do not exclusively breastfed. These problems of breastfeeding usually happen due to limited access to health information about harmful effects in wider community. Mother-in-laws are influential people in the family, including them in breastfeeding education in addition to mothers may improve children's health status and survival.

Objectives: To evaluate effects of breastfeeding education interventions on breastfeeding practices in rural South Ethiopia.

Methods: Community-based, cluster randomized controlled trial, using three-arms parallel group design will be conducted among 510 pregnant women who will be enrolled between the end of first trimester and early second trimester (<16 weeks) of pregnancy. The three arms are: mother alone, mother with mother-in-law and control arm (routine care). The study include 51 non-adjacent clusters (kebeles) for the three arms. This helps minimize information contamination. We implement a simple randomization technique to allocate interventions and control clusters. Interventions will be given at home in eight phases: six times during pregnancy (monthly starting from 4th month up to 9th month), and two times after delivery (within one week and last week of third month). The outcomes are pre-lacteal feeding, colostrum feeding, early initiation and exclusive breastfeeding.

DETAILED DESCRIPTION:
Globally, breastfeeding is recognized as one of the most effective strategies to ensure child health and survival, especially in low and middle-income countries, including Ethiopia, where breast milk substitutes are not always feasible. This is because breast milk is safe, clean, and contains antibodies that help protect against many common childhood illnesses such as acute respiratory infections and diarrheal diseases. In addition, breast milk contains both macro and micro-nutrients that provide nutritional needs, especially in the first six months, and later through complementary foods.

The World Health Organization (WHO) and United Nations Children's Fund (UNICEF) recommend that children initiate breastfeeding within the first hour of birth and be exclusively breastfed for the first 6 months of life, meaning no other foods or liquids are provided, including water.

In Ethiopia, there is a good culture of breastfeeding for a longer duration, as 76% of mothers breastfed their child for at least 2 years, and the median duration of breastfeeding was 23.9 months. However, contrary to the recommendations, still sizeable proportion (41%) of infants do not exclusively breastfeed, 27-36% do not initiate breastfeeding early, 25-46% give pre-lacteal foods/fluids such as butter, honey, and plain water. The first breast milk (colostrum) is also commonly avoided (19-77%) until it is partly or fully removed through manual expression. According to the most recent UNICEF report, the proportion of infants who do not exclusively breastfeed and initiate breastfeeding timely (within 1 hour) were 39% and 77%, respectively. These problems of breastfeeding usually happen due to limited access to health information about harmful effects in the wider community.

Studies reported that, among other factors, poor knowledge of mothers and absence of breastfeeding counseling were significantly associated with poor breastfeeding practices. This suggests that there is a need to increase knowledge through health education to improve breastfeeding practices.

The World Health Assembly (WHA) has set a target to increase the exclusive breastfeeding rate to 50% by 2025. WHO actively promotes breastfeeding as the best source of nourishment for infants and young children, and is working to achieve this target. Ethiopia has made commitments and achieved the target, as the country reached a 59% exclusive breastfeeding rate in 2019. The progress must continue so that all children are able to thrive and the country achieves global targets set by the United Nations, the Sustainable Development Goals (goal 3), to reduce neonatal and child mortalities. Nutrition during pregnancy and childhood is one of Ethiopia's government priority areas, and one of the strategies for child survival is to promote good practices of breastfeeding during the early life of the neonate and good complementary feeding thereafter.

Although pregnancy and childbirth are unique features of women and their contribution is paramount, recognizing the importance of influential peoples in the families such as the husband/partner and mother-in-law is crucial for effective implementations of child health services such as breastfeeding. The husband/partner is an influential person in the family in making decisions about health care in general. In Ethiopia, the mother-in-laws are the most influential people in the family, even they influence more than a husband, especially in breastfeeding practices such as pre-lacteal feeding, colostrum avoidance behavior, and exclusive breastfeeding. They are the one who give the pre-lacteal foods, manually discard colostrum, and push mothers to give foods and fluids for newborns. Mothers, especially young, usually listen and accept the suggestions from mother-in-laws, as they judged as experienced women in pregnancy and childbirth related issues, including feeding newborns and rearing children. In Ethiopia, women usually receive routine maternal and child health care services, while influential peoples such as husband and mother-in-law are commonly overlooked and not involved in the educational services. Previous interventional studies that involved husbands in maternal and child health services education found that men's involvement has a positive impact on improving the utilization of the services. Likewise, previous interventional study conducted in Ethiopia via involving influential peoples in the community (Women Development Army (WAD) leaders found to improve early initiation of breastfeeding and exclusive breastfeeding practices. However, there is a scarcity of evidence that reports the effect of breastfeeding education interventions of mothers and mother-in-laws on improving good practices of breastfeeding in Ethiopia, where people with various socio-cultural characteristics and breastfeeding cultures exist. This is relevant for decision-making in a broader context and to decrease economic losses related to poor practices of breastfeeding, such as household expenditures for treatment and breast milk substitutes when the child gets sick, loss of productive time by parents for caring sick child, and burden on the health care system.

Therefore, this study will provide useful evidence for the implementation of good breastfeeding practices to enhance child health and survival.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are in between the end of their first trimester and the early second trimester (<16 weeks) of pregnancy
* Pregnant women who have not given birth before (nullipara)
* Pregnant women who will give consent
* Pregnant women who have resided in the study area for at least six months.

Exclusion Criteria:

* Pregnant women with previous history of stillbirth
* Pregnant women whose mother-in-law died or unavailable
* Pregnant women who already received breastfeeding practice education intervention from previous trials

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Pre-lacteal feeding | Pre-lacteal feeding will be ascertained in the first week of delivery.
  Pre-lacteal feeding is any fluid given to a child before breastfeeding starts. It can be honey, water, butter, etc. that can be given before newborn starts breastfeeding. In this study, the incidence of pre-lacteal feeding will be assessed by dividing the number of newborns who received pre-lacteal food/fluids to total number of live births. The data will be collected by asking mothers using a face-to-face interview questionnaire.
Colostrum feeding | First week of delivery.
  Colostrum is the first form of breastmilk that is released by the mammary glands after giving birth. It's nutrient-dense and high in antibodies and antioxidants to build a newborn baby's immune system. It changes to breast milk within two to four days after the baby is born. In this study, the incidence of colostrum feeding will be assessed by dividing the number of newborns who feed colostrum to the number of total live births. The data will be collected by asking mothers about whether they give colostrum to the newborn baby or not, using a face-to-face interview questionnaire.
Early initiation of breastfeeding | in this study, early initiation of breastfeeding will be ascertained in the first week of delivery
  Early initiation of breastfeeding is breastfeeding a newborn within one hour of birth. It protects the newborn from acquiring infection and reduces newborn mortality. It facilitates emotional bonding of the mother and the baby and has a positive impact on duration of exclusive breastfeeding. In this study, the incidence of early initiation of breastfeeding will be assessed by dividing the number of newborns who initiated breastfeeding within one hour of birth to the number of total live births. The data will be collected by asking mothers whether they breast fed the newborn within one hour or not, using a face-to-face interview questionnaire.
Exclusive breastfeeding | In this study, exclusive breastfeeding will be evaluated within one week after six months.
  Exclusive breastfeeding means that the infant receives only breast milk. No other liquids or solids are given - not even water - with the exception of oral rehydration solution, or drops/syrups of vitamins, minerals or medicines. In this study, the incidence of exclusive breastfeeding will be assessed by dividing the number of newborns who fed breast milk for up to six months to total number of newborns. The data will be collected by asking mothers using a face-to-face interview questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Belayneh H Jena, PhD, Principal Investigator — Wachemo University

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared for anyone. In this study, the participants data will be used for the analysis purpose only, which will be managed by the principal investigator.

REFERENCES:
- [Result] Infant and Young Child Feeding: Model Chapter for Textbooks for Medical Students and Allied Health Professionals. Geneva: World Health Organization; 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK148965/ PMID 23905206
- [Result] Takele WW, Tariku A, Wagnew F, Ekubagewargies DT, Getinet W, Derseh L, Anlay DZ. Magnitude of prelacteal feeding practice and its association with place of birth in Ethiopia: a systematic review and meta-analysis, 2017. Arch Public Health. 2018 Oct 22;76:63. doi: 10.1186/s13690-018-0308-y. eCollection 2018. PMID 30377528
- [Result] Gebretsadik GG, Tkuwab H, Berhe K, Mulugeta A, Mohammed H, Gebremariam A. Early initiation of breastfeeding, colostrum avoidance, and their associated factors among mothers with under one year old children in rural pastoralist communities of Afar, Northeast Ethiopia: a cross sectional study. BMC Pregnancy Childbirth. 2020 Aug 5;20(1):448. doi: 10.1186/s12884-020-03151-z. PMID 32758166
- [Result] Temesgen H, Negesse A, Woyraw W, Getaneh T, Yigizaw M. Prelacteal feeding and associated factors in Ethiopia: systematic review and meta-analysis. Int Breastfeed J. 2018 Nov 28;13:49. doi: 10.1186/s13006-018-0193-6. eCollection 2018. PMID 30505338
- [Result] Mose A, Dheresa M, Mengistie B, Wassihun B, Abebe H. Colostrum avoidance practice and associated factors among mothers of children aged less than six months in Bure District, Amhara Region, North West, Ethiopia: A community-based cross-sectional study. PLoS One. 2021 Jan 29;16(1):e0245233. doi: 10.1371/journal.pone.0245233. eCollection 2021. PMID 33513154
- [Result] Tsegaye D, Tamiru D, Belachew T. Effect of a theory-based nutrition education intervention during pregnancy through male partner involvement on newborns' birth weights in Southwest Ethiopia. A three-arm community based Quasi-Experimental study. PLoS One. 2023 Jan 17;18(1):e0280545. doi: 10.1371/journal.pone.0280545. eCollection 2023. PMID 36649344
- [Result] Abdulahi M, Fretheim A, Argaw A, Magnus JH. Breastfeeding Education and Support to Improve Early Initiation and Exclusive Breastfeeding Practices and Infant Growth: A Cluster Randomized Controlled Trial from a Rural Ethiopian Setting. Nutrients. 2021 Apr 6;13(4):1204. doi: 10.3390/nu13041204. PMID 33917366
- [Result] Hemming K, Girling AJ, Sitch AJ, Marsh J, Lilford RJ. Sample size calculations for cluster randomised controlled trials with a fixed number of clusters. BMC Med Res Methodol. 2011 Jun 30;11:102. doi: 10.1186/1471-2288-11-102. PMID 21718530
- [Derived] Jena BH, Gemecho TL, Turuse EA, Kebede BA, Adem ZA, Melaku LM, Gelaye KA. Effects of breastfeeding education interventions during pregnancy on breastfeeding practices in rural South Ethiopia: a protocol for cluster randomized controlled trial. BMC Pregnancy Childbirth. 2025 Nov 17;25(1):1224. doi: 10.1186/s12884-025-08290-9. PMID 41249976
- See also: Ethiopia Demographic and Health Survey 2016 — https://dhsprogram.com/publications/publication-fr328-dhs-final-reports.cfm
- See also: Training-of-trainers-manual-for-counseling-on-maternal-infant-and-young-child-nutrition — https://www.iycn.org/resource/ethiopia-training-of-trainers-manual-for-counseling-on-maternal-infant-and-young-child-nutrition/